CLINICAL TRIAL: NCT05820568
Title: Effects and Mechanisms of Change of Two Different Treatments Targeting Worry in Generalised Anxiety Disorder: Study 1 - IU Pilot
Brief Title: Internet Delivered Cognitive Behavior Therapy Based on Intolerance of Uncertainty
Acronym: ORIGAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Forsell, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02380-01-Pilot
Record Dates: First submitted 2022-12-08; First posted 2023-04-19 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: internet delivered treatment; digital mental health services; psychiatry; cognitive behavior therapy; intolerance of uncertainty
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receiving ICBT-IU
  Interventions: Behavioral: ICBT-IU

INTERVENTIONS:
Behavioral: ICBT-IU — Internet delivered Cognitive Behavior Therapy for Generalized Anxiety Disorder based on the Intolerance of uncertainty model of worry

SUMMARY:
The goal of this clinical is to pilot test an internet delivered cognitive behavior therapy (ICBT) based on intolerance of uncertainty (one of several existing specific cognitive models for how worry works) in treating generalised anxiety disorder (GAD). The main aims is to:

* Test the preliminary effect of the intervention in lowering symptoms of GAD as measured by the self report scale GAD-7
* Test procedures for recruitment, assessment, treatment and follow up
* Test the acceptability of the intervention as measured by the Client Satisfaction questionnaire-8, dropout and adverse events

Participants will apply for treatment in an online system, be assessed via video by a licensed clinical psychologist and then receive a 10 week long ICBT intervention based on the intolerance of uncertainty model. This is a pilot study for an upcoming randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more.
* Diagnosis of GAD based on clinical assessment.
* At least 10 points on GAD-7 at screening.
* Proficient in written Swedish.
* Access to internet enabled device and Swedish BankID for authentication
* Able to make sufficient time for the 10 week long treatment
* Consents to study

Exclusion Criteria:

* In need of treatment for other psychiatric diagnosis as priority (eg depression, psychosis) or high risk of suicide based on clinical assessment
* Ongoing risk use of alcohol or drugs
* Ongoing serious somatic of social disease/problem that is deemed to be to much of a hindrance for the completion of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7-item (GAD7) | 10 weeks after treatment start
  Symptoms of generalized anxiety disorder measured by the self report measure GAD7. Scores range from 0-21 with higher scores indicating more generalized anxiety

SECONDARY OUTCOMES:
Treatment credibility | 2 weeks into treatment
  A version of the credibility expectancy questionnaire used at the Internet Psychiatry Clinic in Sweden. Scores range from 5 to 50 with higher scores indicating more credibility.
Satisfaction with treatment | 10 weeks after treatment start
  Client Satisfaction Questionnaire 8 item version (CSQ8). Scores range from 8 to 32; scores of 8-13 indicate poor satisfaction, 14-19 fair satisfaction, 20-25 good satisfaction, and 26-32 excellent satisfaction.
Symptoms of depression including suicidal ideation | 10 weeks after treatment start
  Measured with the Montgomery Åsberg Depression Rating Scale- Self report (MADRS-S). Scores range from 0-54 with higher scores indicating more depression
Intolerance of uncertainty | 10 weeks after treatment start
  Measured with the Intolerance of Uncertainty Scale short version (IUS-12). Scores range from 12-60 with higher scores indicating more intolerance of uncertainty.
Excessive worry | 10 weeks after treatment start
  Measured with the Penn State Worry Questionnaore (PSWQ). Scores range from 16-80 points with more points indicating more worry
Symptoms of depression | 10 weeks after treatment start
  Measured with the Patient Health Questionnaire-9 item self report measure (PHQ9).The scale range is 0-27 with higher scores indication more depression.
WHO Disability Assessment Schedule (WHODAS 2.0) self report (12 items) | 10 weeks after treatment start
  A health and disability metric developed by WHO. Scores range from 0-100% and represent the level of disability with 100% being complete disability to function in everyday life.

OTHER OUTCOMES:
Rate of treatment dropout | 10 weeks after treatment start
  Patient terminates treatment ahead of schedule
Adherence | 10 weeks after treatment start
  Number of modules completed

CONTACTS AND LOCATIONS:
Locations (1):
- Internet Psychiatry Clinic, Psychiatry Southwest, SLSO, Region Stockholm, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No